CLINICAL TRIAL: NCT00595517
Title: A Long Term Study to Investigate the Efficacy and Safety Study of D961H (Esomeprazole) (20 mg Once Daily) for the Prevention of Gastric and/or Duodenal Ulcers Associated With Daily Nonsteroidal Anti-inflammatory Drug (NSAID) Use
Brief Title: Long Term Study to Investigate the Efficacy & Safety of D961H (Esomeprazole) for the Prevention of NSAIDs-induced Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D961HC00005
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-08

CONDITIONS: Gastric Ulcer; Duodenal Ulcer; Rheumatoid Arthritis; Osteoarthritis; Lumbago
Keywords: gastrointestinal; GI; NSAID; Japan; Japanese; Gastric ulcer; duodenal ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Arthritis, Rheumatoid; Osteoarthritis; Low Back Pain | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esomeprazole 20 mg (Experimental): Esomeprazole 20 mg once daily
  Interventions: Drug: Esomeprazole 20 mg

INTERVENTIONS:
Drug: Esomeprazole 20 mg — Esomeprazole 20 mg once daily

SUMMARY:
The purpose of this study is to assess the Safety and tolerability of D961H (Esomeprazole) 20 mg once daily for up to 52 weeks of treatment involving patients with a history of gastric and/or duodenal ulcers receiving daily nonsteroidal anti-inflammatory drug (NSAID) therapy by evaluating AE, clinical laboratory value and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Medical history of gastric and/or duodenal ulcer
* A diagnosis of a chronic condition (rheumatoid arthritis, osteoarthritis, lumbago,etc) that requires daily NSAID use,at least 20 years of age

Exclusion Criteria:

* Having gastric or duodenal ulcer in active or healing stage according to the Sakita/Miwa classification
* History of esophageal, gastric or duodenal surgery
* Having severe liver disease or chronic renal disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naotsugu Oyama, Study Director — AstraZeneca
Locations (3):
- Japan (3):
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Tokyo

REFERENCES:
- [Derived] Sugano K, Kinoshita Y, Miwa H, Takeuchi T; Esomeprazole NSAID Preventive Study Group. Safety and efficacy of long-term esomeprazole 20 mg in Japanese patients with a history of peptic ulcer receiving daily non-steroidal anti-inflammatory drugs. BMC Gastroenterol. 2013 Mar 26;13:54. doi: 10.1186/1471-230X-13-54. PMID 23530709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled 2 Oct 07. Last completed 8 Sept 09. 395 enrolled, 130 registered in study. All registered were included in Full Analysis set and safety analysis set. FAS used for summaries of baseline characteristics and efficacy, safety analysis set for summaries of safety variables.
Pre-assignment Details: Out of 395 enrolled participants, 130 participants were registered and 265 participants were not registered. The major reasons of no registration were 'Incorrect enrollment' (247 participants) and 'Voluntary discontinuation by participant' (18 participants).
Groups:
- Esomeprazole 20mg: Esomeprazole 20 mg once daily oral
Period: Overall Study
Arm/Group | Esomeprazole 20mg
Started | 130
Completed | 111
Not Completed | 19
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 2
Not completed — Recurrence of ulcer | 5
Not completed — usage of prohibited treatment | 1
Not completed — No intention to attend regularly | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esomeprazole 20mg
Number analyzed (Participants) | 130
Age, Customized [Number; unit: Participants]
  < 65 years | 63 [63 to NA]
  65 - 74 years | 43 [43 to NA]
  >= 75 years | 24 [24 to NA]
Sex/Gender, Customized [Number; unit: Participants]
  Male | 35 [35 to NA]
  Female | 95 [95 to NA]

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Without Gastric and/or Duodenal Ulcer up to 4 Weeks After Treatment
Time Frame: up to 4 weeks after treatment
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg
Number analyzed (Participants) | 130
Participants | 130 [NA to NA]

2. Secondary Outcome: Number of Participants Without Gastric and/or Duodenal Ulcer up to 12 Weeks After Treatment
Time Frame: up to 12 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Esomeprazole 20mg
Number analyzed (Participants) | 130
participants | 127 [NA to NA]

3. Secondary Outcome: Number of Participants Without Gastric and/or Duodenal Ulcer up to 24 Weeks After Treatment
Time Frame: up to 24 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Esomeprazole 20mg
Number analyzed (Participants) | 130
participants | 126 [NA to NA]

4. Primary Outcome: Number of Participants Without Gastric and/or Duodenal Ulcer Throughout the Treatment Period
Time Frame: up to 52 weeks
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg
Number analyzed (Participants) | 130
Participants | 125

ADVERSE EVENTS:
Arm/Group | Esomeprazole 20mg
Serious Adverse Events (participants affected / at risk) | 14/130
Other Adverse Events (participants affected / at risk) | 123/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20mg (N=130)
Rheumatoid Arthritis Aggravated (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis Deterioration (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Pyelonephritis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Campylobacter Intestinal Infection (Infections and infestations) | 1
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebral Infarction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20mg (N=130)
Nasopharyngitis (Infections and infestations) | 38
Abdominal Pain Upper (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 11
Stomach Discomfort (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 17
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Contusion (Injury, poisoning and procedural complications) | 7
Headache (Nervous system disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 7
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.